CLINICAL TRIAL: NCT02545803
Title: The Effect of High Frequency Percussive Ventilation on Cerebral Tissue Oxygenation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hasselt University (Other)
Collaborators: Ziekenhuis Oost-Limburg (Other)
Responsible Party: Principal Investigator, prof. dr. Frank Jans, prof. dr., Hasselt University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: VDR4_ZOL1
Record Dates: First submitted 2015-08-20; First posted 2015-09-10 (Estimated); Last update posted 2018-03-27 (Actual); Status verified 2018-03

CONDITIONS: Patients at the Intensive Care Unit (ICU)
MeSH Terms: interventions — Spectroscopy, Near-Infrared

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- study group (Other): Adult patients (age ≥ 18 years) at the Intensive Care Unit (ICU) who become refractory to conventional mechanical ventilation and are switched to HFPV.
  Interventions: Device: Near-Infrared Spectroscopy (NIRS)

INTERVENTIONS:
Device: Near-Infrared Spectroscopy (NIRS) — Near infrared spectroscopy (NIRS) is a non-invasive technique that uses near infrared light between 700 and 1100nm which penetrates several centimeters through skin and bone structures. Light is absorbed by chromophores. There are multiple chromophores which can be detected in the NIR spectrum such as water, lipids, melanin, myoglobin, oxygenated hemoglobin and deoxygenated hemoglobin. Each chromophore has a specific absorption spectrum. By using different wavelengths, it is possible to differentiate chromophores. The difference between oxygenated hemoglobin and deoxygenated hemoglobin can be calculated using the modified Beer-Lambert law, resulting in a numeric value which is a representation of the regional cerebral oxygen saturation

SUMMARY:
Hypoxemia is commonly reported in patients admitted to the Intensive Care Unit (ICU) and may result from acute lung injury/acute respiratory distress syndrome (ALI/ARDS), sepsis, trauma and postoperative complications. In an attempt to preserve or increase the oxygenation, conventional mechanical ventilation is initiated in these patients. Unfortunately, patients frequently become refractory to standard ventilatory techniques and as such, gas exchange remains unaltered or becomes worse. High Frequency Percussive Ventilation (HFPV), on the other hand, is an advanced mode of ventilation which can be a salvage option in these patient cohorts as it has already been proven to improve gas exchange with success. The volumetric diffusive respirator (VDR-4; Percussionary, Corp., Sandpoint, ID) is the only commercially available system to deliver HFPV. This ventilator mechanically ventilates the lung by administering small successive subtidal volumes or percussions at unconventional high frequencies to reach an optimal diffusive oxygenation.

Since it has been known that hypoxemia due to a reduced oxygenation results in secondary brain injury, it is conceivable that the cerebral tissue oxygenation might be impaired as well. It has been strongly suggested that a cerebral tissue oxygenation in the optimal range has an ameliorative influence on hypoxic events and in turn leads to a better clinical outcome. Thus far, no studies have been conducted to investigate if an improved oxygenation by means of a switch to HFPV automatically leads to an increment in the cerebral tissue oxygenation. With the use of Near-Infrared Spectroscopy (NIRS) technology, investigators will investigate whether this alternation of ventilation strategy is associated with a (beneficial) change of the cerebral tissue oxygenation.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age ≥ 18 years) at the Intensive Care Unit (ICU) who become refractory to conventional mechanical ventilation and are switched to HFPV.

Exclusion Criteria:

* Age < 18 years
* Patients with COPD (chronic obstructive pulmonary disease)
* Patients with asthma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-05; Primary Completion 2018-05 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
The association between HFPV and cerebral oxygen saturation | Two hours before switch to HFPV until 24 hours after the switch to HFPV
  The primary objective is to investigate whether a switch from conventional mechanical ventilation to High Frequency Percussive Ventilation is associated with a change of the SctO2. Therefore, a comparison of SctO2-values two hours before and four hours after the switch will be made.

CONTACTS AND LOCATIONS:
Overall Officials: Frank Jans, prof. dr., Principal Investigator — Ziekenhuis Oost-Limburg, Hasselt University
Locations (1):
- Ziekenhuis Oost-Limburg, Genk, Belgium